CLINICAL TRIAL: NCT00535288
Title: A Multicenter, Randomized, Parallel-Group, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Four Different Doses of Org 50081 in the Treatment of Moderate to Severe Vasomotor Symptoms Associated With the Menopause
Brief Title: Dose-Finding Safety and Efficacy Trial of Org 50081 (Esmirtazapine) in the Treatment of Vasomotor Symptoms (177001/P06472/MK-8265-013)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P06472; White Moonstone (Other: Organon Protocol Name); 177001 (Other: Organon Protocol Number)
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Results first posted 2014-07-30 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Postmenopausal Symptoms; Menopause; Vasomotor Symptoms
MeSH Terms: interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Participants receive encapsulated tablets, orally, once daily (QD) for up to 12 weeks.
  Interventions: Drug: Placebo
- Esmirtazapine 2.25 mg (Experimental): Participants receive esmirtazapine, 2.25 mg, encapsulated tablets, orally QD for up to 12 weeks.
  Interventions: Drug: Esmirtazapine
- Esmirtazapine 4.5 mg (Experimental): Participants receive esmirtazapine, 4.5 mg, encapsulated tablets, orally QD for up to 12 weeks.
  Interventions: Drug: Esmirtazapine
- Esmirtazapine 9 mg (Experimental): Participants receive esmirtazapine, 9 mg, encapsulated tablets, orally QD for up to 12 weeks.
  Interventions: Drug: Esmirtazapine
- Esmirtazapine 18 mg (Experimental): Participants receive esmirtazapine, 18 mg, encapsulated tablets, orally QD for up to 12 weeks.
  Interventions: Drug: Esmirtazapine

INTERVENTIONS:
Drug: Esmirtazapine — Four different doses (2.25, 4.5, 9.0, and 18 mg) encapsulated esmirtazapine tablets in Swedish Orange hard gelatin DB-B capsules for blinding purposes. Encapsulated tablets were administered orally once daily in the evening prior to sleep for 12 weeks.
  Other Names: Esmirtazapine maleate; SCH 900265; Org 50081
  Arms: Esmirtazapine 18 mg; Esmirtazapine 2.25 mg; Esmirtazapine 4.5 mg; Esmirtazapine 9 mg
Drug: Placebo — Encapsulated placebo tablets in Swedish Orange hard gelatin DB-B capsules for blinding purposes. Encapsulated tablets were administered orally once daily in the evening prior to sleep for 12 weeks.
  Arms: Placebo

SUMMARY:
To investigate efficacy and safety of 4 doses of esmirtazapine, compared to placebo, in the treatment of moderate to severe hot flushes (vasomotor symptoms) associated with the menopause. Co-primary efficacy endpoints are the frequency and severity of hot flushes after 4 and 12 weeks as compared to Baseline.

DETAILED DESCRIPTION:
The most direct treatment of hot flushes may be by means of 5-HT2A receptor antagonist. Mirtazapine is a potent blocker of 5-HT2A receptors and was found to be effective in reducing the number and intensity of hot flushes in preliminary trials. Also several Selective Serotonin Reuptake Inhibitors (SSRIs) and other similar compounds have been investigated to manage hot flushes, confirming the role of the serotonergic system. In the present trial, the efficacy and safety of four different doses of esmirtazapine compared to placebo were investigated in women with moderate to severe vasomotor symptoms associated with the menopause. The primary objective of this trial was to demonstrate superior efficacy in at least one of the four doses of esmirtazapine as compared to placebo on the four following co-primary endpoints: 1) the mean change from baseline in average daily frequency of moderate and severe vasomotor symptoms at Week 4; 2) the mean change from baseline in average daily frequency of moderate and severe vasomotor symptoms at Week 12; 3) the mean change from baseline in average daily severity of moderate and severe vasomotor symptoms at Week 4; 4) the mean change from baseline in average daily severity of moderate and severe vasomotor symptoms at Week 12. The number and severity of hot flushes was recorded by means of electronic diary by the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women, defined as:

  * 12 months of spontaneous amenorrhea;
  * OR 6 months of spontaneous amenorrhea with serum Follicle Stimulating Hormone (FSH) levels >40 mIU/mL;
  * OR 6 weeks post surgical bilateral oophorectomy with or without hysterectomy.
* Be ≥ 40 and ≤ 65 years of age;
* Have a body mass index (BMI) ≥ 18 and ≤ 32 kg/m^2;
* Minimum of 7 moderate to severe hot flushes per day or 50 per week, as quantified from daily diary recordings during at least 7 days preceding randomization to trial medication;
* Able to handle the electronic diary device after training and having at least 80% compliance on complete daily diary entries during the period prior to randomization;
* Give voluntary written Informed Consent (IC) after the scope and nature of the investigation had been explained, before screening evaluations.

Exclusion Criteria:

* History or presence of any malignancy, except non-melanoma skin cancers;
* Any clinically unstable or uncontrolled renal, hepatic, endocrine, respiratory, hematological, neurological, cardiovascular or cerebrovascular disease that would put the subject at safety risk or mask measure of efficacy;
* History of seizures or epilepsy;
* History or presence of clinically significant depression or other psychiatric disorder which, in the opinion of the investigator, might compromise or confound the subject's participation in the trial;
* Abnormal clinically relevant vaginal bleeding;
* Any clinically relevant (opinion of investigator) abnormal finding during physical, gynecological and breast examination at screening;
* Abnormal, clinically significant results of mammography;
* Abnormal cervical smear test results (corresponding to Pap III and higher, including Low-Grade Squamous Intraepithelial Lesion (LSIL), High-Grade Squamous Intraepithelial Lesion (HSIL), Cervical Intraepithelial Neoplasia (CIN) 1 and higher);
* Hematological or biochemical values at screening outside the reference ranges considered clinically relevant in the opinion of the investigator;
* High Blood Pressure (BP);
* Use of any drug product containing estrogens, progestins, androgens or tibolone prior to screening (and up to and including randomization) within a pre-specified period;
* Any of the following treatments within the last 4 weeks prior to screening (and up to and including randomization):

  * tricyclic antidepressants, Serotonin Noradrenergic Reuptake Inhibitors (SNRIs), SSRIs, Monoamine Oxidase (MAO)-inhibitors, mirtazapine
  * antianxiety drugs, antipsychotics
  * coumarin-derivatives
  * α-adrenergic agents
  * β-blockers
  * dopamine agonists/antagonists
  * opiates, barbiturates
  * raloxifene
  * homeopathic menopausal preparations or other preparations intended to treat climacteric or Central Nervous System (CNS) symptoms
  * hepatic microsomal enzyme-inducing drugs or drugs known to affect or interfere with the pharmacokinetics of mirtazapine;
* Any condition or disease that could affect or interfere with the pharmacokinetics of mirtazapine;
* Subjects sensitive to trial medication or its components;
* Use of any investigational drug and/or participation in another clinical trial within the last eight weeks prior to screening;
* History of alcohol and/or drug abuse within the last two years prior to screening.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 946 (Actual)
Dates: Start 2004-09-15 (Actual); Primary Completion 2006-01-15 (Actual); Study Completion 2006-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Birkhaeuser M, Bitzer J, Braat S, Ramos Y. Esmirtazapine treatment of postmenopausal vasomotor symptoms: two randomized controlled trials. Climacteric. 2019 Jun;22(3):312-322. doi: 10.1080/13697137.2018.1561664. Epub 2019 Feb 4. PMID 30712391
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P06472&kw=P06472&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 946 participants were randomly assigned in this study, however, one participant assigned to placebo never received treatment and one participant assigned to placebo actually received esmirtazapine 18 mg and is included in that group for all study analyses.
Period: Overall Study
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18 mg
Started | 314 (2 participants randomized to receive placebo did not receive placebo) | 162 | 160 | 151 | 158 (One participant randomized to receive placebo received esmirtazapine 18 mg.)
Completed | 260 | 130 | 127 | 122 | 116
Not Completed | 54 | 32 | 33 | 29 | 42
Not completed — Adverse Event | 20 | 19 | 25 | 20 | 30
Not completed — Lost to Follow-up | 0 | 3 | 0 | 0 | 0
Not completed — Lack of Efficacy | 26 | 3 | 4 | 4 | 7
Not completed — Unwilling to cooperate | 6 | 6 | 3 | 3 | 4
Not completed — Other | 2 | 1 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants receive encapsulated tablets, orally, QD for up to 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18 mg | Total
Number analyzed (Participants) | 314 | 162 | 160 | 151 | 158 | 945
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.5 (4.9) | 53.8 (5.0) | 53.7 (4.8) | 54.7 (4.6) | 53.5 (4.7) | 53.8 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 314 | 162 | 160 | 151 | 158 | 945
  Male | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Daily Frequency of Moderate/Severe Vasomotor Symptoms (Frequency Score A) at Week 4
Description: Participants recorded the frequency (number) of vasomotor symptoms (hot flushes) on an electronic diary card (LogPad®) on a daily basis during screening and treatment. Frequency Score A was based on the number of moderate hot flushes + the number of severe hot flushes in one day. Baseline average was derived from, at most, 7 completely observed pre-treatment days. Weekly averages during treatment were calculated if at least 4 days with non-missing data were completely observed; if less than 4 days were completely observed, the averages of the previous week were carried forward (last observation carried forward, or LOCF). If the number of days observed in Week 1 were not sufficient, baseline values were carried forward.
Time Frame: Baseline and Week 4
Population: The Intent-to-Treat (ITT) population, defined as all randomized participants who had at least one pre-baseline and at least one post-baseline average of the number of hot flushes in a week.
Measure: Mean (Standard Deviation); unit: Events per day
Groups:
- Esmirtazapine 18 mg: Participants receive esmirtazapine, 18 mg, encapsulated tablets, orally, QD for up to 12 weeks
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18 mg
Number analyzed (Participants) | 283 | 146 | 144 | 134 | 138
Events per day
  Baseline | 12.1 (5.1) | 12.2 (5.1) | 12.6 (4.7) | 12.3 (4.4) | 11.5 (4.7)
  Week 4 | -3.8 (4.5) | -5.1 (4.1) | -5.7 (4.8) | -5.3 (3.8) | -5.6 (4.4)
Statistical Analysis 1: Comparison: Placebo vs Esmirtazapine 2.25 mg; Test type: Superiority or Other; p < 0.01, ANCOVA — Confidence intervals and p-values were adjusted by (2-sided) Dunnett many-to-one comparison at 0.05 overall Type 1 error rate; Factors for treatment group and (pooled) center and a covariate for the baseline frequency; Difference between least squares means = -1.2, 95% CI 2-sided [-2.2 to -0.2]
Statistical Analysis 2: Comparison: Placebo vs Esmirtazapine 4.5 mg; Test type: Superiority or Other; p < 0.01, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Factors for treatment group and (pooled) center and a covariate for the baseline frequency; Difference between least squares means = -1.7, 95% CI 2-sided [-2.7 to -0.7]
Statistical Analysis 3: Comparison: Placebo vs Esmirtazapine 9 mg; Test type: Superiority or Other; p < 0.01, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Factors for treatment group and (pooled) center and a covariate for the baseline frequency; Difference between least squares means = -1.4, 95% CI 2-sided [-2.4 to -0.4]
Statistical Analysis 4: Comparison: Placebo vs Esmirtazapine 18 mg; Test type: Superiority or Other; p < 0.01, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Factors for treatment group and (pooled) center and a covariate for the baseline frequency; Difference between least squares means = -1.9, 95% CI 2-sided [-2.9 to -0.9]

2. Primary Outcome: Change From Baseline in Average Daily Severity of Moderate/Severe Vasomotor Symptoms (Severity Score A) at Week 4
Description: Participants recorded the severity of hot flushes on a LogPad on a daily basis during screening and treatment. The severity of hot flushes was defined as: mild (sensation of heat without sweating); moderate (sensation of heat with sweating, able to continue activity); and severe (sensation of heat with sweating, causing cessation of activity). Severity Score A was calculated as the number of moderate hot flushes x 2 + the number of severe hot flushes x 3, divided by the total number of moderate and severe hot flushes per week. If no hot flushes were experienced, this was to be recorded as 'no sensation of heat'. Baseline values were based on, at most, 7 completely observed pre-treatment days. If less than 4 days were completely observed during treatment, the averages of the previous week were carried forward (LOCF). If the number of days observed in Week 1 were not sufficient, baseline values were carried forward.
Time Frame: Baseline and Week 4
Population: The ITT population, defined as all randomized participants who had at least one pre-baseline and at least one post-baseline average of the number of hot flushes in a week.
Measure: Mean (Standard Deviation); unit: Severity score
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18 mg
Number analyzed (Participants) | 283 | 146 | 144 | 134 | 138
Severity score
  Baseline | 2.45 (0.30) | 2.45 (0.30) | 2.45 (0.32) | 2.46 (0.30) | 2.40 (0.27)
  Week 4 | -0.07 (0.20) | -0.14 (0.23) | -0.13 (0.23) | -0.15 (0.24) | -0.15 (0.23)
Statistical Analysis 1: Comparison: Placebo vs Esmirtazapine 2.25 mg; Test type: Superiority or Other; p < 0.01, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Factors for treatment group and (pooled) center and a covariate for the baseline severity; Difference between least squares means = -0.07, 95% CI 2-sided [-0.12 to -0.01]
Statistical Analysis 2: Comparison: Placebo vs Esmirtazapine 4.5 mg; Test type: Superiority or Other; p = 0.02, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Factors for treatment group and (pooled) center and a covariate for the baseline severity; Difference between least squares means = -0.06, 95% CI 2-sided [-0.11 to -0.01]
Statistical Analysis 3: Comparison: Placebo vs Esmirtazapine 9 mg; Test type: Superiority or Other; p < 0.01, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Factors for treatment group and (pooled) center and a covariate for the baseline severity; Difference between least squares means = -0.07, 95% CI 2-sided [-0.13 to -0.02]
Statistical Analysis 4: Comparison: Placebo vs Esmirtazapine 18 mg; Test type: Superiority or Other; p < 0.01, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Factors for treatment group and (pooled) center and a covariate for the baseline severity; Difference between least squares means = -0.08, 95% CI 2-sided [-0.14 to -0.03]

3. Primary Outcome: Change From Baseline in Average Daily Frequency of Moderate/Severe Vasomotor Symptoms (Frequency Score A) at Week 12
Description: Participants recorded the frequency (number) of vasomotor symptoms (hot flushes) on a LogPad on a daily basis during screening and treatment. Frequency Score A was based on the number of moderate hot flushes + the number of severe hot flushes in one day. Baseline average was derived from, at most, 7 completely observed pre-treatment days. Weekly averages during treatment were calculated if at least 4 days with non-missing data were completely observed; if less than 4 days were completely observed, the averages of the previous week were carried forward (LOCF). If the number of days observed in Week 1 were not sufficient, baseline values were carried forward.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Events per day
Groups:
- Placebo: Participants receive encapsulated tablets, orally, once daily QD for up to 12 weeks.
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18 mg
Number analyzed (Participants) | 283 | 146 | 144 | 134 | 138
Events per day
  Baseline | 12.1 (5.1) | 12.2 (5.1) | 12.6 (4.7) | 12.3 (4.4) | 11.5 (4.7)
  Week 12 | -4.2 (5.3) | -5.2 (4.6) | -6.0 (4.9) | -5.8 (4.3) | -6.0 (4.6)
Statistical Analysis 1: Comparison: Placebo vs Esmirtazapine 2.25 mg; Test type: Superiority or Other; p = 0.08, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Factors for treatment group and (pooled) center and a covariate for the baseline frequency; Difference between least squares means = -1.0, 95% CI 2-sided [-2.1 to 0.1]
Statistical Analysis 2: Comparison: Placebo vs Esmirtazapine 4.5 mg; Test type: Superiority or Other; p < 0.01, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Factors for treatment group and (pooled) center and a covariate for the baseline frequency; Difference between least squares means = -1.6, 95% CI 2-sided [-2.7 to -0.5]
Statistical Analysis 3: Comparison: Placebo vs Esmirtazapine 9 mg; Test type: Superiority or Other; p < 0.01, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Factors for treatment group and (pooled) center and a covariate for the baseline frequency; Difference between least squares means = -1.5, 95% CI 2-sided [-2.7 to -0.4]
Statistical Analysis 4: Comparison: Placebo vs Esmirtazapine 18 mg; Test type: Superiority or Other; p < 0.01, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Factors for treatment group and (pooled) center and a covariate for the baseline frequency; Difference between least squares means = -2.0, 95% CI 2-sided [-3.1 to -0.9]

4. Secondary Outcome: Change From Baseline in Average Daily Frequency of Moderate/Severe Vasomotor Symptoms (Frequency Score A) by Week Excluding Weeks 4 and 12
Description: as for outcome 3
Time Frame: Baseline and Up to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Events per day
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18 mg
Number analyzed (Participants) | 283 | 146 | 144 | 134 | 138
Events per day
  Baseline | 12.10 (5.10) | 12.19 (5.07) | 12.56 (4.66) | 12.30 (4.39) | 11.52 (4.67)
  Week 1 | -2.21 (3.37) | -3.20 (3.35) | -4.08 (3.79) | -3.63 (2.89) | -4.18 (3.83)
  Week 2 | -3.25 (4.08) | -4.72 (3.85) | -5.19 (4.59) | -4.88 (3.24) | -5.39 (3.96)
  Week 3 | -3.71 (4.39) | -4.82 (4.08) | -5.68 (4.74) | -5.13 (3.68) | -5.59 (4.05)
  Week 5 | -3.90 (4.82) | -5.29 (4.28) | -5.83 (4.72) | -5.50 (3.79) | -5.54 (4.48)
  Week 6 | -4.02 (4.90) | -5.41 (4.43) | -5.96 (4.79) | -5.58 (3.89) | -5.62 (4.71)
  Week 7 | -4.11 (4.96) | -5.33 (4.30) | -6.10 (4.87) | -5.69 (4.28) | -5.93 (4.63)
  Week 8 | -4.04 (5.05) | -5.19 (4.49) | -6.14 (4.72) | -5.86 (4.52) | -5.72 (4.36)
  Week 9 | -4.11 (5.18) | -5.15 (4.65) | -6.23 (4.90) | -5.96 (4.39) | -5.95 (4.77)
  Week 10 | -4.11 (5.42) | -5.18 (4.54) | -5.97 (4.79) | -6.00 (4.36) | -6.11 (4.66)
  Week 11 | -4.20 (5.38) | -5.30 (4.65) | -6.03 (4.86) | -5.86 (4.34) | -5.91 (4.57)

5. Secondary Outcome: Change From Baseline in Average Daily Severity of Moderate/Severe Vasomotor Symptoms (Severity Score A) by Week Excluding Weeks 4 and 12
Description: as for outcome 2
Time Frame: Baseline and up to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Severity score
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18 mg
Number analyzed (Participants) | 283 | 146 | 144 | 134 | 138
Severity score
  Baseline | 2.447 (0.301) | 2.451 (0.297) | 2.449 (0.315) | 2.460 (0.296) | 2.400 (0.274)
  Week 1 | -0.045 (0.124) | -0.081 (0.153) | -0.085 (0.151) | -0.085 (0.159) | -0.108 (0.150)
  Week 2 | -0.063 (0.172) | -0.117 (0.199) | -0.111 (0.212) | -0.140 (0.200) | -0.136 (0.178)
  Week 3 | -0.071 (0.195) | -0.133 (0.214) | -0.119 (0.214) | -0.150 (0.200) | -0.137 (0.240)
  Week 5 | -0.080 (0.215) | -0.141 (0.233) | -0.123 (0.227) | -0.154 (0.225) | -0.151 (0.232)
  Week 6 | -0.075 (0.215) | -0.136 (0.246) | -0.127 (0.234) | -0.140 (0.236) | -0.152 (0.245)
  Week 7 | -0.088 (0.233) | -0.144 (0.236) | -0.131 (0.260) | -0.140 (0.253) | -0.144 (0.257)
  Week 8 | -0.082 (0.239) | -0.142 (0.242) | -0.124 (0.270) | -0.139 (0.254) | -0.133 (0.247)
  Week 9 | -0.083 (0.242) | -0.142 (0.257) | -0.137 (0.260) | -0.130 (0.265) | -0.144 (0.246)
  Week 10 | -0.084 (0.255) | -0.147 (0.261) | -0.125 (0.263) | -0.141 (0.258) | -0.162 (0.252)
  Week 11 | -0.078 (0.261) | -0.159 (0.273) | -0.130 (0.273) | -0.124 (0.257) | -0.156 (0.257)

6. Primary Outcome: Change From Baseline in Average Daily Severity of Moderate/Severe Vasomotor Symptoms (Severity Score A) at Week 12
Description: as for outcome 2
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Severity score
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18 mg
Number analyzed (Participants) | 283 | 146 | 144 | 134 | 138
Severity score
  Baseline | 2.45 (0.30) | 2.45 (0.30) | 2.45 (0.32) | 2.46 (0.30) | 2.40 (0.27)
  Week 12 | -0.08 (0.26) | -0.15 (0.27) | -0.13 (0.27) | -0.13 (0.26) | -0.15 (.026)
Statistical Analysis 1: Comparison: Placebo vs Esmirtazapine 2.25 mg; Test type: Superiority or Other; p = 0.07, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Factors for treatment group and (pooled) center and a covariate for the baseline severity; Difference between least squares means = -0.06, 95% CI 2-sided [-0.12 to 0.00]
Statistical Analysis 2: Comparison: Placebo vs Esmirtazapine 4.5 mg; Test type: Superiority or Other; p = 0.24, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Factors for treatment group and (pooled) center and a covariate for the baseline severity; Difference between least squares means = -0.05, 95% CI 2-sided [-0.11 to 0.02]
Statistical Analysis 3: Comparison: Placebo vs Esmirtazapine 9 mg; Test type: Superiority or Other; p = 0.29, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Factors for treatment group and (pooled) center and a covariate for the baseline severity; Difference between least squares means = -0.04, 95% CI 2-sided [-0.11 to 0.02]
Statistical Analysis 4: Comparison: Placebo vs Esmirtazapine 18 mg; Test type: Superiority or Other; p = 0.02, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Factors for treatment group and (pooled) center and a covariate for the baseline severity; Difference between least squares means = -0.07, 95% CI 2-sided [-0.14 to -0.01]

7. Secondary Outcome: Change From Baseline in Average Daily Moderate/Severe Composite Score (Composite Score A) by Week
Description: Composite Score A was calculated as Severity Score A x Frequency Score A.
Time Frame: Baseline and up to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Composite score
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18 mg
Number analyzed (Participants) | 283 | 146 | 144 | 134 | 138
Composite score
  Baseline | 30.19 (15.42) | 30.41 (14.56) | 31.03 (12.98) | 30.40 (11.81) | 27.87 (12.56)
  Week 1 | -5.65 (8.99) | -8.48 (9.10) | -10.28 (9.19) | -9.43 (7.84) | -10.63 (9.63)
  Week 2 | -8.28 (10.93) | -12.32 (10.18) | -12.98 (11.36) | -12.70 (8.75) | -13.54 (9.89)
  Week 3 | -9.46 (11.92) | -12.63 (11.09) | -14.22 (11.88) | -13.39 (9.82) | -13.89 (10.28)
  Week 4 | -9.79 (12.39) | -13.18 (11.29) | -14.42 (11.88) | -13.70 (10.28) | -13.72 (11.38)
  Week 5 | -9.96 (13.19) | -13.65 (11.77) | -14.47 (11.65) | -14.16 (10.09) | -13.72 (11.33)
  Week 6 | -10.22 (13.40) | -13.89 (11.88) | -14.84 (11.92) | -14.24 (10.26) | -13.95 (12.05)
  Week 7 | -10.42 (13.49) | -13.73 (11.66) | -15.11 (12.32) | -14.42 (11.23) | -14.72 (11.87)
  Week 8 | -10.20 (13.71) | -13.31 (11.98) | -15.19 (11.93) | -14.73 (11.56) | -14.08 (11.21)
  Week 9 | -10.30 (14.06) | -13.20 (12.54) | -15.40 (12.18) | -14.93 (11.20) | -14.67 (12.30)
  Week 10 | -10.26 (14.77) | -13.30 (12.34) | -14.76 (12.07) | -15.03 (11.24) | -15.08 (12.09)
  Week 11 | -10.53 (14.73) | -13.58 (12.61) | -14.92 (12.41) | -14.58 (11.28) | 14.57 (11.85)
  Week 12 | -10.42 (14.56) | -13.25 (12.52) | -14.88 (12.49) | -14.36 (11.17) | -14.71 (12.17)

8. Secondary Outcome: Change From Baseline in Average Daily Frequency of Mild to Severe Vasomotor Symptoms (Frequency Score B) by Week
Description: Participants recorded the frequency (number) of vasomotor symptoms (hot flushes) on a LogPad on a daily basis during screening and treatment. Frequency Score B was based on the number of mild hot flushes + the number of moderate hot flushes + the number of severe hot flushes in one day. Baseline average was derived from, at most, 7 completely observed pre-treatment days. Weekly averages during treatment were calculated if at least 4 days with non-missing data were completely observed; if less than 4 days were completely observed, the averages of the previous week were carried forward (LOCF). If the number of days observed in Week 1 were not sufficient, baseline values were carried forward.
Time Frame: Baseline and up to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Events per day
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18 mg
Number analyzed (Participants) | 283 | 146 | 144 | 134 | 138
Events per day
  Baseline | 13.29 (5.35) | 13.48 (5.35) | 13.66 (4.96) | 13.41 (4.61) | 13.00 (6.09)
  Week 1 | -2.22 (3.41) | -3.24 (3.23) | -3.81 (3.33) | -3.57 (2.96) | -4.16 (4.69)
  Week 2 | -3.35 (4.17) | -4.81 (4.03) | -5.19 (4.46) | -4.79 (3.28) | -5.50 (4.75)
  Week 3 | -3.83 (4.46) | -5.05 (4.15) | -5.66 (4.74) | -5.08 (3.72) | -5.79 (4.88)
  Week 4 | -3.97 (4.63) | -5.37 (4.14) | -6.01 (4.80) | -5.38 (3.98) | -5.85 (5.30)
  Week 5 | -4.06 (4.91) | -5.61 (4.46) | -6.13 (4.81) | -5.57 (4.03) | -5.90 (5.31)
  Week 6 | -4.25 (4.86) | -5.82 (4.51) | -6.32 (4.89) | -5.75 (4.11) | -5.89 (5.24)
  Week 7 | -4.27 (4.85) | -5.69 (4.36) | -6.47 (4.89) | -5.90 (4.45) | -6.15 (5.18)
  Week 8 | -4.19 (4.94) | -5.54 (4.50) | -6.51 (4.72) | -6.06 (4.55) | -6.03 (4.73)
  Week 9 | -4.30 (5.06) | -5.47 (4.71) | -6.59 (4.79) | -6.08 (4.51) | -6.26 (5.26)
  Week 10 | -4.29 (5.39) | -5.59 (4.73) | -6.36 (4.81) | -6.18 (4.46) | -6.35 (5.05)
  Week 11 | -4.43 (5.42) | -5.68 (4.83) | -6.45 (4.91) | -6.08 (4.48) | -6.28 (4.98)
  Week 12 | -4.40 (5.44) | -5.63 (4.71) | -6.45 (4.96) | -6.10 (4.48) | -6.32 (4.99)

9. Secondary Outcome: Change From Baseline in Average Daily Severity of Mild to Severe Vasomotor Symptoms (Severity Score B) by Week
Description: Participants recorded the severity of hot flushes on a LogPad on a daily basis during screening and treatment. The severity of hot flushes was defined as: mild (sensation of heat without sweating); moderate (sensation of heat with sweating, able to continue activity); and severe (sensation of heat with sweating, causing cessation of activity). Severity Score B was calculated as the number of mild hot flushes + the number of moderate hot flushes x 2 + the number of severe hot flushes x 3, divided by the total number of all hot flushes per week. If no hot flushes were experienced, this was to be recorded as 'no sensation of heat'. Baseline values were based on, at most, 7 completely observed pre-treatment days. If less than 4 days were completely observed during treatment, the averages of the previous week were carried forward (LOCF). If the number of days observed in Week 1 were not sufficient, baseline values were carried forward.
Time Frame: Baseline and up to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Severity score
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18 mg
Number analyzed (Participants) | 283 | 146 | 144 | 134 | 138
Severity score
  Baseline | 2.332 (0.369) | 2.331 (0.375) | 2.349 (0.373) | 2.350 (0.347) | 2.270 (0.332)
  Week 1 | -0.080 (0.220) | -0.132 (0.246) | -0.167 (0.245) | -0.140 (0.245) | -0.192 (0.273)
  Week 2 | -0.111 (0.291) | -0.210 (0.342) | -0.223 (0.341) | -0.225 (0.341) | -0.250 (0.312)
  Week 3 | -0.121 (0.307) | -0.217 (0.373) | -0.246 (0.400) | -0.240 (0.337) | -0.272 (0.389)
  Week 4 | -0.113 (0.312) | -0.224 (0.409) | -0.240 (0.388) | -0.249 (0.387) | -0.273 (0.411)
  Week 5 | -0.124 (0.354) | -0.234 (0.411) | -0.228 (0.403) | -0.254 (0.368) | -0.266 (0.409)
  Week 6 | -0.121 (0.360) | -0.222 (0.429) | -0.214 (0.386) | -0.245 (0.396) | -0.275 (0.436)
  Week 7 | -0.142 (0.389) | -0.234 (0.433) | -0.232 (0.444) | -0.242 (0.424) | -0.287 (0.460)
  Week 8 | -0.139 (0.408) | -0.251 (0.440) | -0.234 (0.467) | -0.251 (0.447) | -0.273 (0.463)
  Week 9 | -0.136 (0.408) | -0.245 (0.438) | -0.256 (0.454) | -0.256 (0.462) | -0.292 (0.474)
  Week 10 | -0.143 (0.431) | -0.244 (0.452) | -0.257 (0.465) | -0.257 (0.467) | -0.307 (0.460)
  Week 11 | -0.149 (0.439) | -0.260 (0.467) | -0.245 (0.463) | -0.224 (0.459) | -0.308 (0.477)
  Week 12 | -0.152 (0.457) | -0.255 (0.471) | -0.240 (0.465) | -0.210 (0.450) | -0.280 (0.472)

10. Secondary Outcome: Change From Baseline in Average Daily Mild to Severe Composite Symptoms Score (Composite Score B) by Week
Description: Composite Score B was calculated as Severity Score B x Frequency Score B.
Time Frame: Baseline and up to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Composite score
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18 mg
Number analyzed (Participants) | 283 | 146 | 144 | 134 | 138
Composite score
  Baseline | 31.39 (15.37) | 31.70 (14.47) | 32.13 (12.91) | 31.51 (11.80) | 29.35 (13.55)
  Week 1 | -5.66 (8.94) | -8.53 (8.85) | -10.01 (8.60) | -9.37 (7.74) | -10.61 (10.31)
  Week 2 | -8.38 (10.91) | -12.40 (10.12) | -12.98 (11.05) | -12.60 (8.58) | -13.64 (10.46)
  Week 3 | -9.57 (11.88) | -12.86 (10.89) | -14.40 (11.69) | -13.34 (9.69) | -14.09 (10.80)
  Week 4 | -9.93 (12.36) | -13.48 (11.06) | -14.69 (11.89) | -13.75 (10.24) | -14.01 (11.91)
  Week 5 | -10.12 (13.13) | -13.96 (11.65) | 014.78 (11.54) | -14.22 (10.12) | -14.08 (11.82)
  Week 6 | -10.45 (13.24) | -14.29 (11.65) | -15.19 (11.83) | -14.40 (10.30) | -14.21 (12.22)
  Week 7 | -10.58 (13.23) | -14.09 (11.45) | -15.48 (12.16) | -14.63 (11.18) | -14.93 (12.04)
  Week 8 | -10.34 (13.43) | -13.66 (11.73) | -15.56 (11.76) | -14.92 (11.38) | -14.40 (11.18)
  Week 9 | -10.49 (13.78) | -13.53 (12.33) | -15.77 (11.91) | -15.05 (11.09) | -14.98 (12.44)
  Week 10 | -10.44 (14.56) | -13.71 (12.27) | -15.15 (11.92) | -15.21 (11.11) | -15.32 (12.09)
  Week 11 | -10.76 (14.57) | -13.96 (12.53) | -15.34 (12.27) | -14.79 (11.16) | -14.95 (11.95)
  Week 12 | -10.66 (14.44) | -13.66 (12.32) | -15.32 (12.38) | -14.71 (11.11) | -15.04 (12.17)

11. Secondary Outcome: Total Number of Responders by Week
Description: A participant was defined as a (hot flush) responder for a study week if a reduction of at least 50% for average daily frequency of moderate/severe vasomotor symptoms (hot flushes) (Frequency Score A) compared to Baseline was recorded. A study week was taken into account if at least 4 days were completely observed. The last observation was carried forward if there were less than 4 complete days observed. In cases where Week 1 did not have 4 days that were completely observed, the participant was considered a non-responder. An LOCF approach was used.
Time Frame: Up to 12 weeks
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18 mg
Number analyzed (Participants) | 283 | 146 | 144 | 134 | 138
Participants
  Week 1 | 37 | 29 | 35 | 32 | 42
  Week 2 | 56 | 49 | 60 | 48 | 65
  Week 3 | 85 | 53 | 63 | 47 | 72
  Week 4 | 76 | 58 | 70 | 52 | 71
  Week 5 | 76 | 63 | 65 | 56 | 71
  Week 6 | 84 | 67 | 70 | 55 | 69
  Week 7 | 89 | 59 | 72 | 60 | 75
  Week 8 | 93 | 65 | 73 | 66 | 72
  Week 9 | 96 | 67 | 74 | 68 | 75
  Week 10 | 97 | 65 | 73 | 67 | 77
  Week 11 | 95 | 70 | 78 | 65 | 72
  Week 12 | 99 | 70 | 75 | 65 | 77

12. Secondary Outcome: Total Number of Remitters by Week
Description: A participant was defined as a (hot flush) remitter for a study week if at most one moderate/severe vasomotor symptom per day on average was recorded. A study week was taken into account if at least 4 days were completely observed. The last observation was carried forward if there were less than 4 complete days observed. In cases where Week 1 did not have 4 days that were completely observed, the participant was considered a non-remitter.
Time Frame: Up to 12 weeks
Population: The ITT population, defined as all randomized participants who had at least one pre-baseline and at least one post-baseline average of the number of hot flushes in a week. An LOCF approach was used.
Measure: Number; unit: Participants
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18 mg
Number analyzed (Participants) | 283 | 146 | 144 | 134 | 138
Participants
  Week 1 | 3 | 2 | 7 | 2 | 2
  Week 2 | 6 | 11 | 13 | 8 | 13
  Week 3 | 8 | 15 | 16 | 7 | 17
  Week 4 | 10 | 15 | 18 | 15 | 17
  Week 5 | 13 | 18 | 16 | 12 | 17
  Week 6 | 15 | 15 | 21 | 13 | 18
  Week 7 | 19 | 19 | 22 | 16 | 21
  Week 8 | 23 | 19 | 25 | 18 | 21
  Week 9 | 24 | 19 | 25 | 19 | 26
  Week 10 | 25 | 19 | 25 | 23 | 25
  Week 11 | 25 | 22 | 23 | 21 | 28
  Week 12 | 27 | 23 | 24 | 20 | 26

13. Secondary Outcome: Change From Baseline in Women's Health Questionnaire (WHQ) Sleep Problems Symptoms Domain Score at Week 12
Description: The WHQ is a 36-item, user-friendly, and rapid way of assessing nine domains of physical and emotional health for mid-aged women. Participants self-administered the WHQ questionnaire; scoring is based on a 4-point scale as follows: 'Yes definitely=1', 'Yes sometimes=2', 'No not much=3' and 'No not at all=4'. Each score is transformed to a value '1' for scores '1' and '2' and to a value '0' for scores '3' and '4'. Sleep problems encompass Items 1, 11, and 29 of the 36 total items. The transformed sums of items 1, 11, and 29 were divided by 3 to get the score; therefore, the domain ranges from 0 to 1, where lower values are better.
Time Frame: Baseline and Week 12
Population: All participants who received study drug and had valid answers recorded for the WHQ domain for sleep problems.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Esmirtazapine 9 mg: Participants receive esmirtazapine, 9 mg, encapsulated tablets, orally, QD for up to 12 weeks
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18 mg
Number analyzed (Participants) | 265 | 138 | 134 | 128 | 128
Score on a scale
  Baseline | 0.714 (0.291) [-0.19 to -0.03] | 0.659 (0.321) [-0.18 to 0.01] | 0.684 (0.298) [-0.14 to -0.03] | 0.688 (0.270) | 0.693 (0.260) [-0.20 to -0.03]
  Week 12 | -0.140 (0.325) | -0.232 (0.338) | -0.251 (0.336) | -0.224 (0.381) | -0.195 (0.328)

14. Secondary Outcome: Change From Baseline in WHQ Vasomotor Symptoms Domain Score at Week 12
Description: The WHQ is a 36-item, user-friendly, and rapid way of assessing nine domains of physical and emotional health for mid-aged women. Participants self-administered the WHQ questionnaire; scoring is based on a 4-point scale as follows: 'Yes definitely=1', 'Yes sometimes=2', 'No not much=3' and 'No not at all=4'. Each score is transformed to a value '1' for scores '1' and '2' and to a value '0' for scores '3' and '4'. Vasomotor symptoms encompass Items 19 and 27 of the 36 total items. The transformed sums of items 19+27 are divided by 2 to get the score; therefore, the domain ranges from 0 to 1, where lower values are better.
Time Frame: Baseline and Week 12
Population: All participants who received study drug and had valid answers recorded for the WHQ domain for vasomotor symptoms.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Esmirtazapine 18mg: Participants receive esmirtazapine, 18 mg, encapsulated tablets, orally QD for up to 12 weeks.
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmirtazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18mg
Number analyzed (Participants) | 265 | 138 | 134 | 128 | 128
Score on a scale
  Baseline | 0.983 (0.091) [-0.19 to -0.03] | 0.989 (0.0873) [-0.12 to 0.03] | 0.993 (0.061) [-0.16 to -0.02] | 0.984 (0.087) | 0.984 (0.087) [-0.23 to -0.09]
  Week 12 | -0.085 (0.260) | -0.196 (0.349) | -0.224 (0.381) | -0.117 (0.277) | -0.164 (0.314)

ADVERSE EVENTS:
Time Frame: Non-serious adverse events were collected up to 7 days after the last dose of study drug; serious adverse events were collected for up to 30 days after the last dose of study drug.
Groups:
- Esmertazapine 4.5 mg: Participants receive esmirtazapine, 4.5 mg, encapsulated tablets, orally QD for up to 12 weeks.
Arm/Group | Placebo | Esmirtazapine 2.25 mg | Esmertazapine 4.5 mg | Esmirtazapine 9 mg | Esmirtazapine 18 mg
Serious Adverse Events (participants affected / at risk) | 2/314 | 1/162 | 1/160 | 3/151 | 1/158
Other Adverse Events (participants affected / at risk) | 91/314 | 71/162 | 70/160 | 58/151 | 80/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=314) | Esmirtazapine 2.25 mg (N=162) | Esmertazapine 4.5 mg (N=160) | Esmirtazapine 9 mg (N=151) | Esmirtazapine 18 mg (N=158)
Wolff-Parkinson-White Syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=314) | Esmirtazapine 2.25 mg (N=162) | Esmertazapine 4.5 mg (N=160) | Esmirtazapine 9 mg (N=151) | Esmirtazapine 18 mg (N=158)
Abdominal distension (Gastrointestinal disorders) | 5 (5) | 2 (3) | 3 (3) | 4 (5) | 10 (11)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 8 (9) | 7 (7) | 12 (12) | 9 (10)
Fatigue (General disorders) | 9 (10) | 16 (18) | 26 (28) | 16 (19) | 23 (25)
Oedema peripheral (General disorders) | 3 (4) | 9 (10) | 8 (10) | 3 (6) | 6 (11)
Influenza (Infections and infestations) | 15 (15) | 9 (9) | 3 (3) | 6 (6) | 2 (2)
Weight increased (Investigations) | 6 (6) | 7 (7) | 13 (13) | 11 (11) | 18 (18)
Increased appetite (Metabolism and nutrition disorders) | 4 (4) | 8 (8) | 8 (8) | 10 (11) | 14 (14)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (20) | 6 (6) | 4 (5) | 3 (3) | 6 (6)
Dizziness (Nervous system disorders) | 12 (12) | 8 (8) | 4 (4) | 5 (5) | 13 (14)
Headache (Nervous system disorders) | 33 (52) | 14 (18) | 9 (11) | 5 (14) | 13 (17)
Somnolence (Nervous system disorders) | 6 (7) | 19 (25) | 21 (23) | 11 (12) | 27 (30)
Menopausal symptoms (Reproductive system and breast disorders) | 8 (8) | 5 (5) | 10 (10) | 6 (6) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less